CLINICAL TRIAL: NCT02813525
Title: Ultrasound Monitoring of Fetuses With Vascular Intra-uterine Growth Restriction (IUGR) Using the Isthmus Systolic Index (ISI): Feasibility, Comparison to Normal Fetuses and Association With Perinatal Mortality
Acronym: f-ISI-RCIU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/16
Record Dates: First submitted 2016-06-15; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: IUGR
Keywords: Aortic Isthmus; Isthmic Systolic Index; feasibility; reproducibility; mortality; delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IUGR group: estimated fetal weight <10th percentile associated with an abnormal umbilical artery Doppler with IP>95th percentile or a confirmation of placental vascular disease by histological examination
  Interventions: Other: ISI index on Doppler systolic flow in the aortic isthmus
- CONTROL group: non IUGR fetuses for gestational age (normal for weight, Doppler, and structural analyse)
  Interventions: Other: ISI index on Doppler systolic flow in the aortic isthmus

INTERVENTIONS:
Other: ISI index on Doppler systolic flow in the aortic isthmus — Measure of the ISI index on Doppler systolic flow in the aortic isthmus in the follow-up by ultrasound of the fetus

SUMMARY:
Fetuses with IUGR, there is a correlation between Doppler indices of cardiovascular function and perinatal mortality. An index of systolic flow velocities at the aortic isthmus (ISI) has previously been described in a population of normal fetuses. Fetuses with IUGR, the velocities recorded in the aortic isthmus could be affected and the normal development of the ISI should be changed, because of the increase in placental resistance on one hand, and the gradual deterioration ventricular functions on the other one. Investigators hypothesize that the ISI index in the context of placental insufficiency could provide additional arguments on the extraction timing, the prognosis and the fetal extraction mode to severe hypoxia. The primary outcome of the study is to evaluate in an exploratory manner the feasibility and the potential interest of longitudinal monitoring of fetuses with IUGR by Doppler systolic isthmus and the calculation of the ISI index.

DETAILED DESCRIPTION:
Today evaluating the hemodynamic tolerance of the fetus with IUGR, is based on clinical evidence of fetal well-being and ultrasound arguments, since we know in fact that there is a correlation between Doppler indices of cardiovascular function and perinatal mortality.

The flow to the systolic aortic isthmus may be a marker of systolic performance balance of both ventricles. An index of systolic flow velocities (ISI) has previously been described in a population of normal fetuses. Fetuses with IUGR, the velocities recorded in the aortic isthmus could be affected and the normal development of the ISI should be changed, because of the increase in placental resistance on one hand, and the gradual deterioration ventricular functions on the other one. Investigators hypothesize that the ISI index in the context of placental insufficiency could provide additional arguments on the extraction timing, the prognosis and the fetal extraction mode to severe hypoxia.

The strategy evaluates the feasibility of measuring the ISI index on Doppler systolic flow in the aortic isthmus in the follow-up by ultrasound of the fetus with IUGR due to placental insufficiency.

The ISI is obtained from this flow by calculating the ratio of the minimum systolic velocity (called Nadir) on the peak systolic velocity (called Peak) or Nadir / Peak. The fetal extraction decision (birth) will be taken, blinded the outcome of the ISI, following the protocol of national recommendations for the management of fetuses with IUGR.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age determined by ultrasound dating of the first quarter
* IUGR group: estimated fetal weight <10th percentile associated with

  * An abnormal umbilical artery Doppler with pulsatility index >95th percentile
  * OR a confirmation of placental vascular disease by histological examination
* CONTROL group: non IUGR fetuses for gestational age (normal for weight, Doppler, and structural analyse)

Exclusion Criteria:

* Twin or multiple pregnancy,
* Fetal weight> 10th percentile
* Presence of fetal infection
* Structural fetal anomaly or fetal chromosomal abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vascular IURG fetuses and patients with non-IUGR fetuses.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Compare the evolution of the values of the ISI in the fetus with IUGR relative to those of fetuses without IUGR fetuses for the same gestational age | Up to 3 months

SECONDARY OUTCOMES:
Assess the feasibility of the Doppler and the measure of the parameter | Up to 3 months
  * Obtaining of the sagittal cup or the cross-functional cup of the aortic arch (conformity : yes/no, obtaining: very easy, easy, little easy, difficult, very difficult, impossible).
  * Positioning of the shooting doppler: very easy, easy, little easy, difficult, very difficult, impossible.
  * Doppler flow for the isthmus: conformity yes/no.
  * ISI Measure : very easy, easy, little easy, difficult, very difficult, impossible·
  * Time necessary to obtain the measure (including obtaining of the cup of the aortic arch in sagittal or cross-functional and the measure of the velocities on the Doppler flow).
Compare the reproducibility of the measurement between sonographers with different levels of expertise | Up to 3 months
Estimate the association between ISI index and perinatal mortality and the performance of the ISI in predicting perinatal mortality | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Service de gynécologie-obstétrique et de médecine fœtale, Bordeaux, France